CLINICAL TRIAL: NCT01967342
Title: Reducing Disparities With Literacy-Adapted Psychosocial Treatments for Chronic Pain: A Comparative Trial
Brief Title: Literacy-Adapted Psychosocial Treatments for Chronic Pain --- "Learning About Mastering/My Pain"
Acronym: LAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Whatley Health Services (Unknown); East Carolina University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-021-ME; Easygrants 941 (Other Grant/Funding Number: PCORI (Patient-Centered Outcomes Research Institute))
Record Dates: First submitted 2013-10-16; First posted 2013-10-22 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-03

CONDITIONS: Chronic Pain; Pain; Widespread Chronic Pain; Chronic Pain Syndrome; Chronic Pain Due to Injury
Keywords: chronic pain; pain; chronic pain syndrome; widespread chronic pain; back pain; literacy; health literacy; group therapy; psychosocial treatment; cognitive-behavioral therapy; pain education; health disparities; patient-centered outcomes
MeSH Terms: conditions — Chronic Pain; Pain; Back Pain; Literacy | interventions — Cognitive Behavioral Therapy; Standard of Care; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pain Ed (Experimental): Pain Education: A psychosocial treatment group focusing on providing core pain education to low-income patients who may not have received this information due to existing barriers that often includes limited health literacy. This condition also included medical treatment as usual.
  Interventions: Behavioral: Pain Ed; Other: Usual Care
- CBT for Pain (Experimental): Cognitive-Behavioral Therapy for Pain: A psychosocial treatment group focusing on providing core pain education and cognitive-behavior skills to low-income patients who may not have received this information due to existing barriers that often includes limited health literacy. This condition also included medical treatment as usual.
  Interventions: Behavioral: CBT for Pain; Other: Usual Care
- Usual Care (Active Comparator): Usual Care (Medical Treatment-as-Usual: A control/comparison condition in which patients receive on-going standard care at the federally qualified health center partnering in this research. Facets of care may include medication, surgery, chiropractic, and physical therapy, among others, which are available to all patients in all arms.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Pain Ed — A 10-week psychosocial group treatment for chronic pain that focuses on providing information about the development, course, and treatment of chronic pain, as well as information about factors associated with reduced pain (e.g., sleep). In particular, it seeks to empower patients to take ownership of their chronic pain care through building deeper knowledge about their pain condition and their interactions with the health care system.
  Other Names: EDU; Pain Education; Group Pain Education; Chronic Pain Education; Group Chronic Pain Education
  Arms: Pain Ed
Behavioral: CBT for Pain — A 10-week psychosocial group treatment for chronic pain that focuses on providing information and skills about the development, course, and treatment of chronic pain, as well as information about factors associated with reduced pain (e.g., sleep). In particular, it seeks to empower patients to self-manage their chronic pain through building deeper knowledge about and better skills for improving their pain condition and their interactions with the health care system.
  Other Names: Cognitive-Behavioral Therapy for Pain; Group CBT for Pain; Group Cognitive-Behavioral Therapy for Pain; CBT for Chronic Pain; Group CBT for Chronic Pain; Cognitive-Behavioral Therapy for Chronic Pain; Group Cognitive-Behavioral Therapy for Chronic Pain
  Arms: CBT for Pain
Other: Usual Care — A comparison condition in which patients receive standard individualized medical care from the federally qualified health center partnering on this study. Care can include basic biological interventions, such as medication or surgery, as well as supplementary care such as chiropractic or physical therapy. However, cost has a pragmatic influence on the amount of services provided, sought, and received.
  Other Names: UC; Standard Care; Treatment as Usual; TAU; Medical Treatment as Usual

SUMMARY:
Chronic pain is a significant public health problem that affects over 116 million Americans, costs $600 billion annually, and is unequally borne by people in low-income brackets, especially ethnic minorities. Many individuals also have health literacy deficits (difficulty understanding their illness and difficulty navigating the health care system for treatment) putting them at a greater disadvantage. Treatment usually relies on expensive medical interventions that often have negative side-effects. Psychosocial treatments, like Pain Education and Cognitive-Behavioral Therapy (CBT), show promise, but are usually unavailable. Clinicians are poorly equipped to provide psychosocial treatments to patients with low health literacy. CBT has not been adapted and supported for use in individuals with low health literacy, and even educational materials are often poorly adapted for their needs.

To address this problem, the PI completed a small trial showing benefits from health literacy-adapted pain education and CBT groups for chronic pain in a population with low income and low health literacy. Patients in both treatments reported lower pain by the end of treatment, and the effects were maintained at one year. Patients in the CBT group also reported less depression. The current study uses a larger sample, and directly compares these psychosocial treatments to medical treatment-as-usual to seek better evidence for or against their widespread use in community settings.

Our research questions:

1. In people with chronic pain and low income and/or low literacy, does participating in a health-literacy-adapted psychosocial treatment improve their pain and interference in daily activities due to pain by the end of treatment when compared with a group receiving typical medical care, and are these effects maintained 6 months later?
2. Does participation in the CBT pain management group improve symptoms of depression better than a pain education group by the end of treatment, and are these effects maintained 6 months later?

In partnership with a federally qualified health center, we will enroll 294 patients with chronic pain. Main outcomes will be patient-reported pain intensity, pain interference, depression, and perceived change. From an earlier trial, we expect that our participants will be ~75% female and ~70% African American, and will have low literacy and low income (~60% in the low 15% nationally on word reading, and 90% at or below the poverty threshold).

DETAILED DESCRIPTION:
Study Description

Chronic pain is a major public health problem that is compounded by a number of health-related disparities. Low health literacy presents a notable access barrier to effective treatment as it produces cumulative education and communication deficits. Standard care employs biomedical approaches that are expensive, often invasive, and limited in accessibility and long-term effectiveness. Psychosocial treatments are efficacious, yet few psychosocial interventions have adequately addressed the significant health literacy barriers that exclude a substantial portion of disadvantaged individuals from the benefits of treatment.

Research Questions:

1. In individuals with chronic pain and low socioeconomic standing who are receiving care at a federally qualified health center in the Southern US, does participating in a health-literacy-adapted psychosocial treatment group improve their self-reported pain intensity and interference in physical functioning by the end of treatment when compared with a group receiving standard medical care, and are these effects maintained 6 months later?
2. In these same individuals, does participation in the CBT pain management group improve depressive symptoms better than a pain education group by the end of treatment, and are these effects maintained 6 months later? The proposed study will build on researcher experience developing and evaluating psychosocial treatments for chronic pain in individuals with low socioeconomic standing (SES) and on strong partnerships with community health centers to evaluate two innovative, health-literacy-adapted psychosocial interventions for chronic pain. Both interventions integrate patient feedback, expert opinion, and qualitative patient data.

DESIGN

We propose a three-group, community-based randomized, controlled, comparative effectiveness trial. Participants will be patients receiving care from a federally qualified primary care clinic. Patients are expected to be mostly ethnic minority females living below the poverty line with significant unmet need for chronic pain treatment. Patients will be randomly assigned by group to a standard medical treatment control, a pain education group, or a cognitive-behavioral therapy group. Primary outcomes are patient-reported pain intensity, pain interference in physical functioning, and psychological symptoms, all highly relevant to patient-provider decision-making.

Aims:

1. Evaluate the feasibility, acceptability, and comparative effectiveness of health literacy-adapted psychosocial group treatments to a standard-treatment control.
2. Evaluate the comparative effectiveness of treatment groups on depressive symptoms, and evaluate all outcomes for heterogeneity of treatment effects.

STUDY IMPACT

* Systems: Produces a new, low-cost treatment option for community health clinics.
* Providers: Offers options for treatments over and above surgery and medication.
* Patients: Provides information to patients on the benefits of psychosocial treatment on outcomes that matter.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 19 yrs-old in order to consent to treatment.
2. Must have received at least one diagnosis consistent with chronic pain by a physician at one of the participating primary care clinics.
3. Must have experienced pain most days of the month for 3 months, and although pain may have more than one pain source, all pain must be non-malignant (e.g., not cancer- or HIV-related).
4. Must be able to speak and understand English.
5. Must have a telephone or other avenue of communication for contact regarding the study.

Exclusion Criteria:

1. Must not demonstrate significant cognitive impairment (based on results of a cognitive screener).
2. Must not have current, uncontrolled serious psychological disturbance (e.g., schizophrenia, bipolar disorder) or active substance abuse (based on responses to a structured diagnostic interview).
3. Must have minimal literacy skills (i.e., read at the 1st grade level).
4. Must have been stabilized for at least 4 weeks on current pain and psychotropic medication regimen to reduce potential confounds to treatment results.
5. Must not have a surgery scheduled for the intervention period (~3 months).
6. Must neither be currently receiving a psychosocial treatment for pain (though they may be receiving psychotherapy for non-pain difficulties) nor be a participant in our previous treatment studies.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2013-09-12 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly E. Thorn, Ph.D., Principal Investigator — University of Alabama at Birmingham; Joshua C. Eyer, Ph.D., Study Director — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - Whatley Health Services, Inc., Tuscaloosa, Alabama
  - University of Alabama, Department of Psychology, Tuscaloosa, Alabama
  - East Carolina University, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The complete data set may be obtained by request from the PI. The dataset will be available in November.

REFERENCES:
- [Background] Thorn BE, Day MA, Burns J, Kuhajda MC, Gaskins SW, Sweeney K, McConley R, Ward CL, Cabbil C. Randomized trial of group cognitive behavioral therapy compared with a pain education control for low-literacy rural people with chronic pain. Pain. 2011 Dec;152(12):2710-2720. doi: 10.1016/j.pain.2011.07.007. Epub 2011 Sep 14. PMID 21920668
- [Background] Day MA, Thorn BE, Kapoor S. A qualitative analysis of a randomized controlled trial comparing a cognitive-behavioral treatment with education. J Pain. 2011 Sep;12(9):941-52. doi: 10.1016/j.jpain.2011.02.354. Epub 2011 Aug 11. PMID 21839689
- [Background] Kuhajda MC, Thorn BE, Gaskins SW, Day MA, Cabbil CM. Literacy and cultural adaptations for cognitive behavioral therapy in a rural pain population. Transl Behav Med. 2011 Jun;1(2):216-23. doi: 10.1007/s13142-011-0026-2. PMID 24073046
- [Background] Day MA, Thorn BE. The relationship of demographic and psychosocial variables to pain-related outcomes in a rural chronic pain population. Pain. 2010 Nov;151(2):467-474. doi: 10.1016/j.pain.2010.08.015. PMID 20817401
- [Background] Campbell LC. Addressing literacy as a barrier in delivery and evaluation of cognitive-behavioral therapy for pain management. Pain. 2011 Dec;152(12):2679-2680. doi: 10.1016/j.pain.2011.09.004. Epub 2011 Sep 29. No abstract available. PMID 21963312
- [Background] Thorn BE, Burns JW. Common and specific treatment mechanisms in psychosocial pain interventions: the need for a new research agenda. Pain. 2011 Apr;152(4):705-706. doi: 10.1016/j.pain.2010.12.017. Epub 2011 Jan 11. No abstract available. PMID 21227586
- [Derived] Burns JW, Gerhart J, Van Dyke BP, Morais CA, Newman AK, Thorn B. Examination of mechanism effects in cognitive behavioral therapy and pain education: analyses of weekly assessments. Pain. 2021 Sep 1;162(9):2446-2455. doi: 10.1097/j.pain.0000000000002237. PMID 34448755
- [Derived] Newman AK, Thorn BE. Intersectional identity approach to chronic pain disparities using latent class analysis. Pain. 2022 Apr 1;163(4):e547-e556. doi: 10.1097/j.pain.0000000000002407. PMID 34252906
- [Derived] Morais CA, Newman AK, Van Dyke BP, Thorn B. The Effect of Literacy-Adapted Psychosocial Treatments on Biomedical and Biopsychosocial Pain Conceptualization. J Pain. 2021 Nov;22(11):1396-1407. doi: 10.1016/j.jpain.2021.04.005. Epub 2021 May 15. PMID 34004347
- [Derived] Newman AK, Morais CA, Van Dyke BP, Thorn BE. An Initial Psychometric Evaluation of the Pain Concepts Questionnaire in a Low-SES Setting. J Pain. 2021 Jan;22(1):57-67. doi: 10.1016/j.jpain.2020.05.002. Epub 2020 Jun 27. PMID 32603873
- [Derived] Van Dyke BP, Newman AK, Morais CA, Burns JW, Eyer JC, Thorn BE. Heterogeneity of Treatment Effects in a Randomized Trial of Literacy-Adapted Group Cognitive-Behavioral Therapy, Pain Psychoeducation, and Usual Medical Care for Multiply Disadvantaged Patients With Chronic Pain. J Pain. 2019 Oct;20(10):1236-1248. doi: 10.1016/j.jpain.2019.04.006. Epub 2019 Apr 22. PMID 31022555
- [Derived] Newman AK, Kapoor S, Thorn BE. Health Care Utilization for Chronic Pain in Low-Income Settings. Pain Med. 2018 Dec 1;19(12):2387-2397. doi: 10.1093/pm/pny119. PMID 29905879
- [Derived] Thorn BE, Eyer JC, Van Dyke BP, Torres CA, Burns JW, Kim M, Newman AK, Campbell LC, Anderson B, Block PR, Bobrow BJ, Brooks R, Burton TT, Cheavens JS, DeMonte CM, DeMonte WD, Edwards CS, Jeong M, Mulla MM, Penn T, Smith LJ, Tucker DH. Literacy-Adapted Cognitive Behavioral Therapy Versus Education for Chronic Pain at Low-Income Clinics: A Randomized Controlled Trial. Ann Intern Med. 2018 Apr 3;168(7):471-480. doi: 10.7326/M17-0972. Epub 2018 Feb 27. PMID 29482213
- [Derived] Newman AK, Van Dyke BP, Torres CA, Baxter JW, Eyer JC, Kapoor S, Thorn BE. The relationship of sociodemographic and psychological variables with chronic pain variables in a low-income population. Pain. 2017 Sep;158(9):1687-1696. doi: 10.1097/j.pain.0000000000000964. PMID 28570481
- See also: The Thorn Pain Management Team Web Site — http://pmt.ua.edu
- See also: Whatley Health Services, Inc. — http://www.whatleyhealth.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Usual Care (Medical Treatment-as-Usual): A control/comparison condition in which patients receive standard individualized medical care from the federally qualified health center partnering on this study. Care can include basic biological interventions, such as medication or surgery, as well as supplementary care such as chiropractic or physical therapy.
- CBT for Pain: Cognitive-Behavioral Therapy for Pain: A 10-week psychosocial group treatment for chronic pain that focuses on providing core pain education and cognitive-behavior skills to low-income patients who may not have received this information due to existing barriers that often includes limited health literacy. In particular, it seeks to empower patients to self-manage their chronic pain through building deeper knowledge about and better skills for improving their pain condition and their interactions with the health care system. Sessions occur once per week for a duration of 1.5 hours.
- Pain Ed: Pain Education: A 10-week psychosocial group treatment for chronic pain that focuses on providing core pain education to low-income patients who may not have received this information due to existing barriers that often includes limited health literacy. In particular, it seeks to empower patients to take ownership of their chronic pain care through building deeper knowledge about their pain condition and their interactions with the health care system. Sessions occur once per week for a duration of 1.5 hours.
Period: Overall Study
Arm/Group | Usual Care | CBT for Pain | Pain Ed
Started | 98 | 95 | 97
5-week Follow-up | 83 | 78 | 76
10-week Follow-up | 78 | 83 | 80
Completed (6-month follow-up) | 71 | 70 | 68
Not Completed | 27 | 25 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | CBT for Pain | Pain Ed | Total
Number analyzed (Participants) | 98 | 95 | 97 | 290
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 96 | 90 | 93 | 279
  >=65 years | 2 | 5 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (8.7) | 52.2 (8.5) | 49.9 (9.2) | 50.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 67 | 69 | 205
  Male | 29 | 28 | 28 | 85
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African-American | 60 | 75 | 59 | 194
  White/Caucasian | 38 | 20 | 38 | 96
Brief Pain Inventory (BPI) Severity [Mean (Standard Deviation); unit: units on a scale] — Pain severity scores were calculated from the mean of four items asking participants to rate the most severe pain, least severe pain, and average pain over the past 7 days, and current pain on an 11-point Likert Scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine). Higher scores indicate greater pain severity.
  units on a scale | 6.5 (1.6) | 6.5 (1.8) | 6.5 (1.5) | 6.5 (1.6)
Brief Pain Inventory (BPI) Interference [Mean (Standard Deviation); unit: units on a scale] — Pain interference scores were calculated from the mean of 7 items asking participants to rate interference due to pain in various domains on an 11-point Likert scale ranging from 0 (no interference) to 10 (complete interference). Higher scores indicate greater pain interference.
  units on a scale | 6.6 (2.1) | 6.7 (2.1) | 6.6 (1.9) | 6.6 (2.0)
Patient Health Questionnaire-9 items (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionaire-9 (PHQ-9) is a 9-item self-report module. Each item is measured on a scale of 0 (not at all) to 3 (nearly every day). Scores can range from 0 to 27. Higher scores indicate greater severity of depressive symptoms.
  units on a scale | 12.8 (6.4) | 11.7 (6.1) | 11.9 (6.8) | 12.1 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory-Intensity (BPI-Intensity)
Description: Brief Pain Inventory-Intensity indicates level of pain intensity. Higher scores (range 0-10) reflect higher perceived pain severity.
Time Frame: Post-treatment (10-weeks) and follow-up (6 months)
Population: The predicted mean estimates were based on latent growth modeling from mplus using all participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | CBT for Pain | Pain Ed
Number analyzed (Participants) | 78 | 82 | 80
units on a scale
  Post-treatment (10-weeks) | 6.19 (1.81) | 5.42 (2.29) | 5.68 (2.04)
  Follow-up (6-months): number analyzed (Participants) | 71 | 69 | 67
  Follow-up (6-months) | 5.95 (1.84) | 5.82 (2.22) | 5.97 (1.99)
Statistical Analysis 1: Comparison: Usual Care; A piecewise linear growth model examined changes in BPI-Intensity within Usual Care between pre-treatment and 10-week post-treatment; Test type: Superiority or Other; p = .165, Mixed Models Analysis; Mean Difference (Net) = -0.268, Standard Error of Mean -0.193
Statistical Analysis 2: Comparison: Usual Care; A piecewise linear growth model examined changes in BPI-Intensity within Usual Care between post-treatment and 6-month follow-up; Test type: Superiority or Other; p = .216, Mixed Models Analysis; Mean Difference (Net) = -0.245, Standard Error of Mean 0.198
Statistical Analysis 3: Comparison: CBT for Pain; A piecewise linear growth model examined changes in BPI-Intensity within CBT group between the pre-treatment and 10-week post-treatment; Test type: Superiority or Other; p < .001, Mixed Models Analysis; Mean Difference (Net) = -1.052, Standard Error of Mean 0.189
Statistical Analysis 4: Comparison: CBT for Pain; A piecewise linear growth model examined changes in BPI-Intensity within CBT group between the post-treatment and 6-month follow-up; Test type: Superiority or Other; p = .070, Mixed Models Analysis; Mean Difference (Net) = 0.361, Standard Error of Mean 0.199
Statistical Analysis 5: Comparison: Pain Ed; A piecewise linear growth model examined changes in BPI-Intensity within Pain Ed group between the pre-treatment and 10-week post-treatment; Test type: Superiority or Other; p < .001, Mixed Models Analysis; Mean Difference (Net) = -0.823, Standard Error of Mean 0.191
Statistical Analysis 6: Comparison: Pain Ed; A piecewise linear growth model examined changes in BPI-Intensity within Pain Ed group between the post-treatment and 6-month follow-up; Test type: Superiority or Other; p = .519, Mixed Models Analysis; Mean Difference (Net) = 0.131, Standard Error of Mean 0.203

2. Secondary Outcome: Brief Pain Inventory-Interference (BPI-Interference)
Description: Brief Pain Inventory-Intensity indicates level of pain interference. Higher scores (range 0-10) reflect higher perceived pain interference.
Time Frame: Post-treatment (10-weeks) and follow-up (6 months)
Population: The predicted mean estimates were based on latent growth modeling from mplus using all participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | CBT for Pain | Pain Ed
Number analyzed (Participants) | 78 | 83 | 80
units on a scale
  10-week post-treatment | 6.11 (2.52) | 5.01 (2.73) | 5.46 (2.43)
  6-month follow-up: number analyzed (Participants) | 71 | 70 | 68
  6-month follow-up | 6.32 (2.18) | 5.55 (2.75) | 5.98 (2.36)
Statistical Analysis 1: Comparison: Usual Care; A piecewise linear growth model examined changes in BPI-Interference within Usual Care group between the pre-treatment and 10-week post-treatment; Test type: Superiority or Other; p = .196, Mixed Models Analysis — To control for multiple comparisons in secondary outcomes, a corrected alpha level was calculated using the Benjamini-Hochberg correction method. Smallest p-value compared to .025; Largest p-value compared to .050; Mean Difference (Net) = -0.310, Standard Error of Mean 0.247
Statistical Analysis 2: Comparison: Usual Care; A piecewise linear growth model examined changes in BPI-Interference within Usual Care group between the post-treatment and 6-month follow-up; Test type: Superiority or Other; p = .447, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.182, Standard Error of Mean 0.239
Statistical Analysis 3: Comparison: CBT for Pain; A piecewise linear growth model examined changes in BPI-Interference within CBT for Pain group between the pre-treatment and 10-week post-treatment; Test type: Superiority or Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.643, Standard Error of Mean 0.241
Statistical Analysis 4: Comparison: CBT for Pain; A piecewise linear growth model examined changes in BPI-Interference within CBT for Pain group between the post-treatment and 6-month follow-up; Test type: Superiority or Other; p = .021, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.548, Standard Error of Mean 0.237
Statistical Analysis 5: Comparison: Pain Ed; A piecewise linear growth model examined changes in BPI-Interference within Pain Ed group between the pre-treatment and 10-week post-treatment; Test type: Superiority or Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.999, Standard Error of Mean 0.244
Statistical Analysis 6: Comparison: Pain Ed; A piecewise linear growth model examined changes in BPI-Interference within Pain Ed group between the post-treatment and 6-month follow-up; Test type: Superiority or Other; p = .305, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.250, Standard Error of Mean 0.243

3. Secondary Outcome: Patient Health Questionnaire - 9 (PHQ-9)
Description: Depressive symptoms were assessed using the Patient Health Questionnaire-9 (PHQ-9; range 0-27; higher scores indicate greater severity).
Time Frame: Post-treatment (10-weeks) and follow-up (6 months)
Population: The predicted mean estimates were based on latent growth modeling from mplus using all participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | CBT for Pain | Pain Ed
Number analyzed (Participants) | 78 | 83 | 80
units on a scale
  Post-treatment (10-weeks) | 11.42 (6.56) | 9.13 (5.77) | 9.59 (6.12)
  Follow-up (6-months): number analyzed (Participants) | 71 | 70 | 68
  Follow-up (6-months) | 11.58 (7.09) | 9.73 (6.70) | 10.53 (6.35)
Statistical Analysis 1: Comparison: Usual Care; A piecewise linear growth model examined changes in PHQ-9 within Usual Care group between the pre-treatment and 10-week post-treatment; Test type: Superiority or Other; p = .082, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.086, Standard Error of Mean 0.623
Statistical Analysis 2: Comparison: Usual Care; A piecewise linear growth model examined changes in PHQ-9 within Usual Care group between the post-treatment and 6-month follow-up; Test type: Superiority or Other; p = .652, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.240, Standard Error of Mean 0.532
Statistical Analysis 3: Comparison: CBT for Pain; A piecewise linear growth model examined changes in PHQ-9 within CBT for Pain group between the pre-treatment and 10-week post-treatment; Test type: Superiority or Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -2.416, Standard Error of Mean 0.612
Statistical Analysis 4: Comparison: CBT for Pain; A piecewise linear growth model examined changes in PHQ-9 within CBT for Pain group between the post-treatment and 6-month follow-up; Test type: Superiority or Other; p = .241, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.619, Standard Error of Mean 0.528
Statistical Analysis 5: Comparison: Pain Ed; A piecewise linear growth model examined changes in PHQ-9 within Pain Ed group between the pre-treatment and 10-week post-treatment; Test type: Superiority or Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -2.251, Standard Error of Mean 0.617
Statistical Analysis 6: Comparison: Pain Ed; A piecewise linear growth model examined changes in PHQ-9 within Pain Ed group between the post-treatment and 6-month follow-up; Test type: Superiority or Other; p = .422, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.434, Standard Error of Mean 0.541

4. Secondary Outcome: Patient Global Impression of Change (PGIC), Pain Intensity
Description: The Patient Global Impression of Change (PGIC) assesses self-perceived changes in pain intensity. Scores were dichotomized such that responses of "very much better" and "much better" were recoded as 1 and all other responses were coded as zero, as performed by Cherkin et al. (2016), in order to indicate clinically meaningful improvement on pain intensity. The following outcome measure data table reports the number of participants per group reporting clinically meaningful improvement at post-treatment (10-weeks) and follow-up (6-months).
Time Frame: Retrospective self-report at post-treatment (10-weeks) and follow-up (6-months).
Population: Only participants who completed the post-treatment (10-weeks) and follow-up (6-months) assessments were included in the following analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | CBT for Pain | Pain Ed
Number analyzed (Participants) | 78 | 82 | 80
Participants
  Post-treatment (10-weeks) | 6 | 33 | 23
  Follow-up (6-months): number analyzed (Participants) | 71 | 69 | 68
  Follow-up (6-months) | 6 | 19 | 22
Statistical Analysis 1: Comparison: Usual Care vs CBT for Pain; Odds ratios were computed to describe the likelihood of participants in each treatment condition reporting clinically meaningful improvement on the PGIC-pain intensity relative to the other groups at post-treatment (6-months); Test type: Superiority or Other; p < .001, Mixed Models Analysis; Odds Ratio (OR) = 8.45 — CBT vs. TAU
Statistical Analysis 2: Comparison: Usual Care vs Pain Ed; Odds ratios were computed to describe the likelihood of participants in each treatment condition reporting clinically meaningful improvement on the PGIC-pain intensity relative to the other groups at post-treatment (10-weeks); Test type: Superiority or Other; p = .001, Mixed Models Analysis; Odds Ratio (OR) = 5.53 — EDU vs. TAU
Statistical Analysis 3: Comparison: CBT for Pain vs Pain Ed; Odds ratios were computed to describe the likelihood of participants in each treatment condition reporting clinically meaningful improvement on the PGIC-pain intensity relative to the other groups at pre-treatment (10-weeks); Test type: Superiority or Other; p = .217, Mixed Models Analysis; Odds Ratio (OR) = 1.53 — CBT vs. EDU
Statistical Analysis 4: Comparison: Usual Care vs CBT for Pain; Odds ratios were computed to describe the likelihood of participants in each treatment condition reporting clinically meaningful improvement on the PGIC-pain intensity relative to the other groups at follow-up (6-months); Test type: Superiority or Other; p = .009, Mixed Models Analysis; Odds Ratio (OR) = 3.81 — CBT vs. TAU
Statistical Analysis 5: Comparison: Usual Care vs Pain Ed; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = .001, Mixed Models Analysis; Odds Ratio (OR) = 5.32 — EDU vs. TAU
Statistical Analysis 6: Comparison: CBT for Pain vs Pain Ed; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = .389, Mixed Models Analysis; Odds Ratio (OR) = 0.72 — CBT vs. EDU

ADVERSE EVENTS:
Time Frame: 2 years, 11 months and 4 days.
Description: Participants completed four assessments over the course of the study. Assessors asked about adverse events at these assessments, using a safety alert form prepared for the trial. Participants in the CBT and EDU conditions also completed weekly measures at the time of the weekly meeting over the 10-week class, and were asked about adverse events on a weekly basis. For each safety alert/adverse event, participants were asked whether it was related to being in the study.
Arm/Group | Usual Care | CBT for Pain | Pain Ed
Serious Adverse Events (participants affected / at risk) | 3/98 | 1/95 | 2/97
Other Adverse Events (participants affected / at risk) | 12/98 | 4/95 | 14/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=98) | CBT for Pain (N=95) | Pain Ed (N=97)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gout flare on right knee and foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal Infection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Unknown reason for hospitalization (General disorders) | 1 (1) | 0 (0) | 0 (0) — ER visit and hospitalization from 10/24/14 to 10/26/14 for unknown cause. Participant reported that this event was unrelated to pain or participation in the study.
Female organ surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=98) | CBT for Pain (N=95) | Pain Ed (N=97)
Musculoskeletal pain exacerbation (Musculoskeletal and connective tissue disorders) | 12 | 4 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes